CLINICAL TRIAL: NCT03621072
Title: AN OPEN-LABEL, RANDOMIZED, SINGLE-DOSE, 2-WAY CROSSOVER BIOEQUIVALENCE STUDY COMPARING FLUCONAZOLE 150 MG CAPSULE (MANUFACTURED AT PFIZER DALIAN, CHINA) WITH FLUCONAZOLE 150 MG CAPSULE (MANUFACTURED AT PFIZER FAREVA, AMBOISE, FRANCE) UNDER FASTED AND FED CONDITIONS IN HEALTHY CHINESE SUBJECTS
Brief Title: Bioequivalence (BE) Study Comparing Fluconazole 150mg Capsule Manufactured in China and in France
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0561025
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Bioequivalence
Keywords: Fluconazole; Bioequivalence; Phase I; Chinese; Healthy Subjects
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, single-dose, 2-way crossover bioequivalence study under fasted and fed conditions in healthy Chinese subjects. Under each condition, subjects will be randomized to one of the 2 treatment sequences. Each treatment sequence will consist of 2 periods, separated by a washout period of at least 14 days between each period. For sequence 1, first localized originator and then originator will be administered. The order for sequence 2 is originator and localized originator.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Reference (Other): Fluconazole 150mg Capsule Originator
  Interventions: Drug: Fluconazole 150mg Capsule Originator
- Experimental (Experimental): Fluconazole 150mg Capsule Localized Originator
  Interventions: Drug: Fluconazole 150mg Capsule Localized Originator

INTERVENTIONS:
Drug: Fluconazole 150mg Capsule Originator — 150mg fluconazole capsule (originator) manufactured at Pfizer Fareva, Amboise, France
  Other Names: The originator, Reference
  Arms: Reference
Drug: Fluconazole 150mg Capsule Localized Originator — 150mg Fluconazole capsule (localized originator) manufactured at Pfizer, Dalian, China
  Other Names: The localized originator, Experimental
  Arms: Experimental

SUMMARY:
China Food and Drug Administration (CFDA) initiated a generic consistency evaluation program to evaluate the quality and efficacy of the products manufactured in China in 2016. This is a bioequivalence study to support the program and to demonstrate the bioequivalence between the 150 mg fluconazole capsule manufactured at Pfizer Dalian, China (the localized originator, Test) and the 150 mg fluconazole capsule manufactured at Pfizer Fareva, Amboise, France (the originator, Reference) in healthy Chinese subjects under fasted and fed conditions. This open-lable, randomized, single-dose 2-way crossover study will enroll approximately 18 subjects for each condition. The primary endpoints are fluconazole area under the plasma concentration-time curve from time zero to 72 hours post-dose (AUC72) and Cmax.

DETAILED DESCRIPTION:
This trial is a bioequivalence study to support a generic consistency evaluation program, initiated by the China Food and Drug Administration (CFDA), for the evaluation of quality and efficacy of the products manufactured in China. The selected strength of 150 mg capsule is the approved highest strength of capsule formulation in China. The 150 mg dose was selected for evaluation in this study as it is one of the commonly used clinically approved doses. The primary objective is to demonstrate the bioequivalence between the 150 mg fluconazole capsule manufactured at Pfizer Dalian, China (the localized originator, Test) and the 150 mg fluconazole capsule manufactured at Pfizer Fareva, Amboise, France (the originator, Reference) administered as a single oral dose in healthy Chinese subjects under fasted and fed conditions. The primary endpoints are fluconazole area under the plasma concentration-time curve from time zero to 72 hours post-dose (AUC72) and peak plasma concentrations (Cmax).

The secondary objective is to evaluate the safety and tolerability of fluconazole administered as a single oral dose of 150 mg capsule manufactured at Pfizer Dalian, China and 150 mg capsule manufactured at Pfizer Fareva, Amboise, France in healthy Chinese subjects under fasted and fed conditions. The secondary endpoint is adverse events (AEs). Other endpoints include time to reach Cmax (Tmax) of fluconazole, safety laboratory tests and vital signs.

In each group, subjects will be randomized to one of the 2 treatment sequences. Each treatment sequence will consist of 2 periods, separated by a washout period of at least 14 days between each period.

On Day 1 of each period in both groups, each subject will be administered investigational product at approximately 8:00 AM (± 2 hours). Blood samples for the analysis of fluconazole in plasma will be collected at pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48 and 72 hours post dose in each period. Vital signs, physical examination, laboratory tests and 12 lead electrocardiogram (ECG) will be performed at specified times. Tolerability and safety will be assessed for all treatments by monitoring AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese male and female subjects, between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate (PR) measurement, 12-lead ECG, or clinical laboratory tests.
2. Body Mass Index (BMI) of 18 to 28 kg/m**2, inclusive; and a total body weight >=50 kg for males and >= 45 kg for females.
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
5. Subjects must be of Chinese ethnicity (individuals currently residing in mainland China who were born in China and have both parents of Chinese descent)

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. A positive urine drug screen.
4. History of regular alcohol consumption exceeding 7 drinks/week for female subjects or 14 drinks/week for male subjects (1 drink = 150 mL of wine or 360 mL of beer or (45 mL of hard liquor) within 6 months of Screening.
5. Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day within 3 months of Screening; a positive urine nicotine test.
6. Treatment with an investigational drug (which has not been approved for registration) within 30 days preceding the first dose of investigational product. If the investigational drug has a long elimination half-life, the washout period will be longer with a recommendation of five elimination half-lives.
7. Screening BP >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility.
8. Screening supine 12 lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS complex >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
9. Female subjects of childbearing potential and fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
10. Female subjects who are breastfeeding or with positive pregnancy test at Screening and during the study period.
11. Use of prescription or nonprescription drugs and dietary supplements within 7 days prior to the first dose of investigational product. If the concomitant medication has a long elimination half-life, the washout period will be longer with a recommendation of five elimination half-lives. As an exception, acetaminophen/paracetamol may be used at doses of <=1 g/day. Limited use of nonprescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.
12. Blood donation (excluding plasma donations) of approximately 400 mL or more within 60 days prior to dosing.
13. History of sensitivity to heparin or heparin induced thrombocytopenia.
14. History of hypersensitivity to fluconazole or any components of its formulation.
15. History of hepatitis B or hepatitis C; positive testing for hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), hepatitis C antibody (HCVAb), treponema pallidum antibody (TPPA) or human immunodeficiency virus (HIV) antibody.
16. Unwilling or unable to comply with the criteria in the Lifestyle Guidelines described in this protocol.
17. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
18. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
AUC0-72 | 0-72 hours
  Area under the plasma concentration-time profile from time zero to 72 hours post dose based on observed plasma concentrations at time points 0 (prior-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6,8, 10, 12, 24, 48 and 72 hours after dose using linear/log trapezoidal methods
Cmax | 0-72hours
  Maximum plasma concentration among observed plasma concentrations at time points 0 (prior-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6,8, 10, 12, 24, 48 and 72 hours after dose

SECONDARY OUTCOMES:
Adverse Events | Day 1 to Day 18 or early termination, plus at least 28 calendar days and up to 35 calendar days after the last administration of the investigational product
  All observed or volunteered safety events regardless of treatment group or suspected causal relationship to the investigational product(s) will be reported during study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Wuxi People's Hospital//Phase One Unit, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Chen N, He Q, Ma Y, Liu S, Wei H, Peng A. Pharmacokinetics and Bioequivalence of Fluconazole Capsules Manufactured in France and China in Healthy Chinese Participants: Open-Label, Randomized, Single-Dose, 2-Way, Crossover Bioequivalence Study Under Fasted and Fed Conditions. Clin Pharmacol Drug Dev. 2023 Jun;12(6):572-578. doi: 10.1002/cpdd.1248. Epub 2023 Apr 10. PMID 37036155
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0561025&StudyName=An+Open-label%2C+Randomized%2C+Single-dose%2C+2-way+Crossover+Bioequivalence+Study+Comparing+Fluconazole+150+Mg+Capsule+%28manufactured+At+Pfizer+Dalian%2C+China%29+With+Fluconazole+150+Mg+Capsule+%28manufactured+At+Pfizer+Fareva%2C+Amboise%2C+France%29+Under+Fasted+And+Fed+Conditions+In+Healthy+Chinese+Subjects